CLINICAL TRIAL: NCT06704425
Title: The Impacts of Chronic Non-specific Low Back Pain on Cognitive Functions of Older Adults: a Cross-sectional Study
Brief Title: The Impacts of Chronic Non-specific Low Back Pain on Cognitive Functions of Older Adults
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Principal Investigator, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20231212006; 1-CD63 (Other Grant/Funding Number: Reserach Center of Smart Aging)
Record Dates: First submitted 2024-07-03; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-08

CONDITIONS: Chronic Non-Specific Low Back Pain; Cognitive Decline; Cross-Sectional Study; Older Adults; Brain Imaging
Keywords: Chronic Non-Specific low back pain; cognitive decline; Cross-Sectional study; older adults; brain imaging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic non-specific low back pain group: Participants with chronic non-specific low back pain (CNSLBP) should have: (1) CNSLBP that has lasted for at least 3 months, typically occurs in the area between the 12th rib to the iliac crest with and without leg pain and without a known pathoanatomical cause; (2) an average pain intensity of ≥ 5 out of 10 on an 11-point numerical rating scale (NRS) in the last 7 days, where 0 means "no pain"and 10 means "worst pain imaginable"; and (3) pain occurring more than 3 days per week.
  Interventions: Other: For observational studies, participants are not assigned an intervention as part of the study.
- Healthy group: Healthy controls should not have CNSLBP in the last 36 months.
  Interventions: Other: For observational studies, participants are not assigned an intervention as part of the study.

INTERVENTIONS:
Other: For observational studies, participants are not assigned an intervention as part of the study. — For observational studies, participants are not assigned an intervention as part of the study.

SUMMARY:
Chronic non-specific low back pain (CNSLBP) is a prevalent condition among older adult and has been associated with an increased risk of executive function impairment. Studies have shown that older adults with chronic pain are more likely to show poor cognitive performance than healthy controls. Cognitive performance is particularly important when managing pain in older adults, especially for some executive functions (e.g., inhibition, switching, working memory) because pain and executive functions have their bidirectional relationship. Further, executive dysfunctions are associated with a decline in functional status among older adults, particularly the impairment of instrumental activities of daily living. Given the above, the preservation of executive functions emerges as a pivotal consideration among old adults with CNSLBP. Studies have provided preliminary evidence of the correlation between brain changes associated with chronic pain and cognitive functions. For example, multisite chronic pain may contribute to an increased risk of cognitive decline via structural change in hippocampal atrophy. For another example, functional brain changes in chronic pain reduced the deactivation of several key default mode network regions, thereby predisposing individuals to cognitive impairments. Despite the aforementioned brain changes, no research has provided direct evidence to support the hypothesis that structural and functional brain changes caused by CNSLBP in older adults may be associated with cognitive decline. Specifically, whether CNSLBP may lead to structural changes (e.g., smaller hippocampal, cerebellar gray matter, white matter volume in the right frontal region) and/or functional changes (e.g., deactivation of default mode network regions, heightened activation in the anterior cingulate cortex) associated with cognitive decline remains unclear. With the help of neuroimaging, the knowledge about the underlying brain mechanisms between CNSLBP (chronic non-specific low back pain) and executive functions can be explained.

To gain a better understanding of the brain mechanisms underlying executive function decline in older adults with CNSLBP, this study will directly compare pain intensity, executive functions, brain structure, and functional changes of the brain between older adults with CNSLBP and age-matched healthy controls. The results of this study have the potential to quantify the association between CNSLBP-related brain changes and executive functions in older adults, and provide insights into the development of new treatment strategies to improve or prevent executive function decline in older adults with CNSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Older adults with and without chronic non-specific low back pain (CNSLBP) aged between 60 and 85 years
* Having normal cognitive function (Hong Kong Montreal Cognitive Assessment ≥ 26)13
* Right-handed
* Cantonese speaking
* Having at least 6 years of formal education and know how to read and write Chinese
* Agreeing to sign an informed consent form
* Being able to communicate via email or text message because several study measures will be collected electronically.

Exclusion Criteria:

* Inability to ambulate without assistance from another person (canes or walkers will be allowed)
* Having specific causes of LBP (e.g., spinal stenosis, lumbar disc herniation, spondylolisthesis, recent vertebral fracture, spinal infection)
* Having other concurrent musculoskeletal conditions at other body parts (e.g., fibromyalgia, or neck or knee pain)
* Self-reported history of lumbar or lower extremity surgery
* Self-reported history of neurological or psychiatric disorders (e.g., stroke, brain surgery, head trauma; schizophrenia, multiple personality disorder, dissociative identity disorder, stroke) or self-reported cancer history
* Self-reported specific inflammatory disorder: rheumatoid arthritis, rheumatica, scleroderma, lupus, or polymyositis
* Unexplained, unintended weight loss of 20 lbs or more in the past year
* Cauda equina syndrome
* Uncorrected visual deficit
* Drug or alcohol addiction
* Taking alcohol, opioids or benzodiazepines medicines 24 hours before the experiment
* Claustrophobia
* Contraindications for undergoing the magnetic resonance imaging (MRI) examination based on the MRI safety screening form of University Research Facility in Behavioral and Systems Neuroscience at The Hong Kong Polytechnic University

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with chronic non-specific low back pain (CNSLBP) should have:
  * CNSLBP that has lasted for at least 3 months, typically occurs in the area between the 12th rib to the iliac crest with and without leg pain and without a known pathoanatomical cause;
  * an average pain intensity of ≥ 5 out of 10 on an 11-point numerical rating scale (NRS) in the last 7 days, where 0 means "no pain" and 10 means "worst pain imaginable"; and
  * pain occurring more than 3 days per week. In addition, healthy controls should not have CNSLBP in the last 36 months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessment | Baseline
  11-point numerical rating scale, ranged from 0 to 10, higher scores indicate higher pain intensity.

SECONDARY OUTCOMES:
Depression, anxiety, and stress test | Baseline
  The Chinese version of the short Depression Anxiety Stress Scales, scores ranged from 0 to 13, higher scores for each domain (depression, anxiety, and stress) indicate more respective problems.
Disability evaluation | Baseline
  The Hong Kong Chinese Version of the Roland-Morris Disability Questionnaire has 24 items. Scores ranged from 0 to 24, higher scores indicate worse disability.
Working memory test inside magnetic resonance imaging scanning | Baseline
  The digit 2-back task, more response accuracy of digits indicates better working memory
Cognitive flexibility test inside magnetic resonance imaging scanning | Baseline
  The More Odd Shifting task, It requires participants to switch between different mental sets or rules, such as identifying odd numbers or shifting between different categories. Better response accuracy indicates better cognitive flexibility
Cognitive inhibition test inside magnetic resonance imaging scanning | Baseline
  Color-Word Matching Stroop Task, more correct matching indicate better ability to inhibit cognitive interference
Perseveration and abstract reasoning test outside magnetic resonance imaging scanning | Baseline
  The Modified Wisconsin Card Sorting Test, more correct matching of cards indicate better perseveration and abstract reasoning.
Working memory Test outside magnetic resonance imaging scanning | Baseline
  The Verbal Digits Forward and Backward Test, more correct recall of digits indicate better working memory and executive function
Cognitive flexibility test outside magnetic resonance imaging scanning | Baseline
  The Trail Making Tests, a neuropsychological test of visual attention and task switching, completing the trail correctly within a shorter period of time means better cognitive flexibility
Inhibition test outside magnetic resonance imaging scanning | Baseline
  Go/NoGo task, more response accuracy indicates better control of inhibition.
Pain catastrophizing assessment | Baseline
  The Chinese version of Pain Catastrophizing Score. The scores ranged from 0 to 13, higher scores indicate more pain catatrophizing thought.
Pain drawing test | Baseline
  The body map scoring system indicates the location of participants' painful site
Frailty status assessment | Baseline
  Fatigue, Resistance, Ambulation, Illness, and Loss, the presence of 3 of 5 item characteristics indicate the presence of frailty, scores ranged from 0 to 5. Lower scores mean more frailty.
Physical activity assessment | Baseline
  Physical Activity Scale for the Elderly; it has 3 domains (leisure, household, and occupation activities) to measure physical activity levels of adults aged 65 or above. higher scores indicate more active.
Sleep quality assessment | Baseline
  Pittsburgh Sleep Quality Index. It has 7 domains to measure sleep quality , sleep latency, sleep duration, habital sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Scores ranged from 0 to 21, higher scores indicate poorer sleep quality.
Cognitive function screening | Baseline
  Hong Kong Montreal Cognitive Assessment. It is a cognitive screening tool specifically adapted for Chinese older adults in Hong Kong. It is designed to detect mild cognitive impairment and dementia. A score < 26 suggests participant has mild cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold YL Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- Hong Kong (3):
  - University Research Facility in Behavioral and Systems Neuroscience, Hong Kong, Hong Kong
  - Arnold YL Wong, Hong Kong, None Selected
  - Department of Rehabilitation Sciences, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided